CLINICAL TRIAL: NCT04439253
Title: MATCH Treatment Subprotocol G: Phase II Study of Crizotinib in Patients With ROS1 Translocations (Other Than Patients With Non-Small Cell Lung Cancer)
Brief Title: Testing Crizotinib as a Potential Targeted Treatment in Cancers With ROS1 Genetic Changes (MATCH-Subprotocol G)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03269; NCI-2020-03269 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-G (Other: ECOG-ACRIN Cancer Research Group); EAY131-G (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (crizotinib) (Experimental): Patients receive crizotinib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Given PO
  Other Names: Alkixen; Crizocent; MET Tyrosine Kinase Inhibitor PF-02341066; PF 02341066; PF-02341066; PF-2341066; PF02341066; Xalkori

SUMMARY:
This phase II MATCH treatment trial identifies the effects of crizotinib in patients whose cancer has a genetic change called ROS1 translocation. Crizotinib may block a protein called ROS1, which may be needed for cancer cell growth. Researchers hope to learn if crizotinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive crizotinib orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must be positive for translocation or inversion events involving the ROS1 gene via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)

Exclusion Criteria:

* Patients must not have NSCLC with ROS1 rearrangements
* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have known hypersensitivity to crizotinib or compounds of similar chemical or biologic composition
* Patients using drugs or foods that are known potent CYP3A4 inhibitors or inducers will be excluded
* Patients must not have had prior therapy with any ROS1 inhibitor including crizotinib, ceritinib, foretinib, cabozantinib, AP26113, ASP3026, WZ-5-126, TAE684, KIST301072, KIST301080, AZD1480, PF-06463922, RXDX-101 and PF-3922

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron S Mansfield, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol G was activated on August 12, 2015. A total of 5 patients were assigned to this arm after screening, 2 from screening cohort and 3 from outside assay. Of the 5 patients, 4 patients were enrolled to arm G between August 2015, and September 2018.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol G, patients had to have an ROS1 translocations (other than patients with non-small cell lung cancer).
Groups:
- Treatment (Crizotinib): Patients receive crizotinib 250 mg PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Crizotinib: Given PO
Period: Overall Study
Arm/Group | Treatment (Crizotinib)
Started (All 4 patients enrolled were eligible and treated in the arm.) | 4
Completed (Treatment continued until disease progression or intolerability.) | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Disease progression | 2
Not completed — Complicating disease | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Treatment (Crizotinib)
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 54 [47 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for the detailed definitions of response criteria. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Crizotinib)
Number analyzed (Participants) | 4
percentage of participants | 25 [1.3 to 75.1]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first.
  Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in NeuroOncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Crizotinib)
Number analyzed (Participants) | 4
percentage of participants | 50 [22 to 100]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Crizotinib)
Number analyzed (Participants) | 4
months | 4.3 [0.53 to NA] — Median PFS 90% CI upper bound could not be determined due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All 4 cases that received protocol treatment were monitored for adverse events.
Arm/Group | Treatment (Crizotinib)
All-Cause Mortality (participants affected / at risk) | 4/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Crizotinib) (N=4)
Abdominal pain (Gastrointestinal disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Crizotinib) (N=4)
Anemia (Blood and lymphatic system disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04439253/Prot_000.pdf